CLINICAL TRIAL: NCT00469118
Title: Clinical Efficacy and Safety of Axiom Worldwide DRX9000 Axial Decompression
Brief Title: Clinical Efficacy and Safety of Axiom Worldwide DRX9000 Axial Decompression System for Treatment of Low Back Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Financial concerns with device manufacturer.
Sponsor: NEMA Research, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Pergolizzi, MD, Principal Investigator, NEMA Research, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AXW01
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRX Treatment (Experimental): 20 treatments of spinal decompression over a six week period. Each session lasts about 45 minutes and consists of a 28-minute treatment on the DRX9000™ machine followed by 15 minutes of cold therapy to the lumbar paravertebral muscles.
  Interventions: Device: DRX9000™
- Conservative Care (No Intervention): Conservative non surgical therapy for 6 weeks prior to beginning DRX9000 treatment

INTERVENTIONS:
Device: DRX9000™ — Nonsurgical spinal decompression
  Arms: DRX Treatment

SUMMARY:
This study will document efficacy and safety of the Axiom Worldwide DRX9000™ for treatment of low back pain (LBP) in a prospective, randomized, crossover, multicenter trial utilizing a standardized clinical research multimodal protocol. During the first two weeks subjects are randomized to receive either conservative care or DRX treatment first and then cross over to receive either conservative care or DRX treatment the next 6 weeks. This study will test the hypothesis that standardized 6-week treatment regimen of spinal decompression using DRX9000™ will reduce chronic lower back pain more than conservative therapy (current baseline therapy).

DETAILED DESCRIPTION:
This study will document efficacy and safety of the Axiom Worldwide DRX9000™ for treatment of low back pain (LBP) in a prospective, randomized, crossover, multicenter trial utilizing a standardized clinical research multimodal protocol. During the first two weeks subjects are randomized to receive either conservative care or DRX treatment first and then cross over to receive either conservative care or DRX treatment the next 6 weeks. This study will test the hypothesis that standardized 6-week treatment regimen of spinal decompression using DRX9000™ will reduce chronic lower back pain more than conservative therapy (current baseline therapy

ELIGIBILITY:
Inclusion Criteria:

* In addition to a diagnosis of LBP, ALL of the following criteria must be met:

  * Male or female, >18 years of age
  * Able to provide written informed consent (ICF) to the IRB approved clinical multimodal protocol
  * Chronic (onset more than 12 weeks) low back pain with an intensity level of > 4 on a verbal rating scale for pain (VRS) of 0-10 (with 0 = no pain and 10 = worst possible pain)
  * Completed necessary diagnostic medical history evaluation forms as described in the protocol to confirm the patient's diagnosis and eligibility for the study
  * Willing and able to complete the 6 week 20 session DRX9000 outpatient treatments and a minimum of 6 months follow-up

Exclusion Criteria:

* If ANY of the following exclusion criteria are present, the subject is NOT eligible:

  * Pregnancy
  * Evidence of neurologic motor deficits on clinical examination
  * Evidence of spinal cord compression, metastatic cancer, tumor, hematoma, infection or compression fracture
  * Severe spinal stenosis
  * Litigation for health-related claim (in process or pending), Worker's Compensation, or Personal Injury cases
  * Previous spine fusion surgery or instrumentation
  * Hemiplegia or paraplegia
  * Significant cardiovascular or metabolic disease, or abdominal aortic aneurysm
  * Unwillingness to postpone other types of therapy for LBP that are not listed as adjuncts in the research protocol
  * Known alcohol abuse or drug abuse
  * Height less than 4 feet 10 inches (147 cm) or greater than 6 feet 8 inches (203 cm)
  * Body weight greater than 300 pounds (136 kg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is lower back pain measured on an 11-point numeric rating scale (VRS) with 0 reflecting no pain at all and 10 the worst imaginable pain. | 1 year

SECONDARY OUTCOMES:
Incidence of adverse events | 1 year
Recurrence rate, measured by the proportion of patients with VRS ≥ 4 | 1 year
Proportion of patients using adjuvant analgesic medication | 1 year
Functional capacity, measured by the established Oswestry Disability Index | 1 year
Patient's satisfaction with procedures and treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joseph V Pergolizzi, MD, Principal Investigator — NEMA Research, Inc.; Charlotte Richmond, PhD, Study Director — NEMA Research, Inc.
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States